CLINICAL TRIAL: NCT01467414
Title: A Trial Investigating the Pharmacodynamic Properties of NN1250 in Japanese Subjects With Type 2 Diabetes
Brief Title: A Trial Investigating the Effect of NN1250 in Japanese Subjects With Type 2 Diabetes
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This trial was terminated due to low recruitment
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN1250-3763; 2011-001850-27 (EudraCT Number); U1111-1120-7444 (Other: WHO)
Record Dates: First submitted 2011-10-31; First posted 2011-11-08 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NN1250 (Experimental)
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Injected s.c. (under the skin) once daily for 6 days

SUMMARY:
This trial is conducted in Europe. The aim of this clinical trial is to investigate the pharmacodynamic (the effect of the investigated drug on the body) properties of NN1250 (insulin degludec) in Japanese subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Japanese subject aged 20-70 years (both inclusive)
* Japanese passport holder
* Japanese-born parents
* Type 2 diabetes mellitus (as diagnosed clinically) for at least 12 months
* Treated with insulin for at least 3 months
* Body Mass Index (BMI) maximum 33.0 kg/m^2
* Glycosylated haemoglobin A1c (HbA1c) maximum 10.0%
* Fasting C-peptide below 1.0 nmol/L

Exclusion Criteria:

* Use of oral antidiabetic drugs (OADs) and/or glucagon like peptide-1 (GLP-1) receptor agonists (exenatide, liraglutide) within 3 months prior to screening
* Subject who has donated any blood or plasma in the past month or more than 500 mL within 3 months prior to screening
* Not able or willing to refrain from smoking and use of nicotine gum or transdermal nicotine patches during the inpatient period
* Supine blood pressure at screening (after resting for 5 min) minimum 180 mmHg for systolic and/or minimum 100 mmHg for diastolic

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Area under the glucose infusion rate curve during one dosing interval at steady state | Within 0-24 hours after last dosing

SECONDARY OUTCOMES:
Maximum glucose infusion rate at steady state | Within 0-24 hours after last dosing
Area under the serum insulin degludec concentration-time curve during one dosing interval at steady state | Within 0-24 hours after last dosing
Maximum observed serum insulin degludec concentration at steady state | Within 0-24 hours after last dosing

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com